CLINICAL TRIAL: NCT00070824
Title: Functional Brain Imaging - Acupuncture and Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R21AT000960-01A1 (NIH)
Record Dates: First submitted 2003-10-08; First posted 2003-10-13 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2007-09

CONDITIONS: Osteoarthritis
Keywords: Acupuncture; SPECT; f-MRI; Functional brain imaging; RCT
MeSH Terms: conditions — Osteoarthritis | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Experimental): Patients with osteoarthritis pain at rest
  Interventions: Procedure: acupuncture
- A (Experimental): Normal Subjects without pain
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture

SUMMARY:
The goal of this study is to use single photon emission computed tomography (SPECT) and functional magnetic resonance imaging (f-MRI) of the brain to study the response of both normal participants and participants with Osteoarthritis (OA) of the knee to acupuncture.

DETAILED DESCRIPTION:
Recent experimental studies in both animal and humans have begun to demonstrate some measurable physiologic effects that are associated with acupuncture, suggesting the possibility of a neurophysiologic explanation. In addition, brain research continues to uncover a complex set of endogenous neurologic control systems, such that it has become clear that the brain plays a major role in the modulation of pain perception and control. If acupuncture can be demonstrated to have a consistent effect on specific areas of the brain, it will become possible to explore the potential efficacy of acupuncture based on measurable neurophysiologic responses.

ELIGIBILITY:
Inclusion criteria:

* Seen in an outpatient clinical setting
* Have active knee OA of >6 months including Kellgren x-ray changes >2 from an x-ray report <12 months old or new x-ray interpretation
* Moderate unilateral only pain (average >4/10 on a 0-10 likert scale) for more than 5 out of 7 days
* Have the capacity to understand the requirements of the study and complete the baseline studies in a reasonable time frame, as determined by the interviewer

Exclusion criteria:

* Having had acupuncture before (must be acupuncture naïve)
* Any history of claustrophobia that could affect the subject's ability to tolerate the f-MRI study
* Hip or ankle disease by history or exam severe enough to cause pain >2/10 daily
* Bleeding disorder or current use of warfarin or heparin by patient history
* Other primary causes of chronic knee pain, per the referring physician, including chondromalacia patella, torn meniscus or ligament injury.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
SPECT Cerebral Bloodflow | 24 hours

SECONDARY OUTCOMES:
0-10 Numeric Rating Scale for Pain Intensity | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: John T. Farrar, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States